CLINICAL TRIAL: NCT03710551
Title: Stool Composition and GI Tolerance in Infants Fed a Term Infant Formula With a New Fat Blend Plus L.Reuteri: a Randomized Controlled Trial
Brief Title: Happy Smooth Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 16.28.INF
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Infant Term Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Infant Formula (Experimental): Experimental Infant Formula with a new fat blend plus L. reuteri
  Interventions: Other: Experimental Infant Formula
- Standard Infant Formula (Active Comparator): Standard bovine milk-based infant formula.
  Interventions: Other: Standard Infant Formula

INTERVENTIONS:
Other: Experimental Infant Formula — Standard bovine milk-based infant formula with a new fat blend plus L. reuteri, fed ad libitum
  Arms: Experimental Infant Formula
Other: Standard Infant Formula — Standard bovine milk-based infant formula, fed ad libitum
  Arms: Standard Infant Formula

SUMMARY:
The purpose of this study is to evaluate the stool composition and GI tolerance of an experimental formula with a new fat blend plus L. reuteri vs control formula.

DETAILED DESCRIPTION:
Double-blind, randomized, controlled clinical trial. The purpose of this study is to evaluate the stool composition and GI tolerance of 140 healthy, term infants fed with an infant formula with a new fat blend plus L. reuteri vs a standard infant formula. All enrolled infants will participate in the trial for approximately 71 days.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Infants whose parents/LAR have reached the legal age of majority in the Philippines
* Infants whose parent(s)/LAR are willing and able to comply with scheduled visits, and the requirements of the study protocol
* Infants whose parent(s)/LAR are able to be contacted directly by telephone throughout the study
* Healthy term, singleton infant at birth
* Between 21 to 28 days post-natal age at enrollment visit
* Weight-for-age ≥ 5th and ≤ 95th percentile according to World Health Organization growth tables/charts
* Infants of parent(s)/LAR who have previously made the decision to formula feed their infant at the time of enrollment

Exclusion Criteria:

* Infants with conditions requiring infant feedings other than those specified in the protocol
* Infants receiving complementary foods or liquids
* Infants who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results
* Infants who are presently receiving or have received medications that could interfere with the interpretation of the study results

Ages: 21 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
Stool Consistency Score | Study Day 57, corresponding to infant age of 78-85 days
  3-day Gastrointestinal (GI) Symptom and Behavior Diary, a parent-reported symptom diary to record stool consistency and stool frequency over the 3 consecutive days.
  A validated 5-point pictorial representation of the consistency of the stool for infants ≤1 year (1=watery, 2=runny, 3=mushy soft, 4=formed, 5=hard) will be provided in the stool diary for parent(s)/LAR to visually assess the infants' stools.
  Stool consistency will be compared between formula groups The baseline stool consistency value will also be included in the model as a covariate.
  the percentage of stools in each category (watery, runny, mushy soft, formed, or hard) will be calculated by visit for each infant and then will be summarized using the appropriate descriptive statistics. Figures composed of a series of histograms will be produced for each 3-day stool diary period.

SECONDARY OUTCOMES:
GI Tolerance | which corresponds to infant age of 21-28, 43-50, and 78-85 days.
  Infant Gastrointestinal Symptom Questionnaire (IGSQ)
  Overall GI symptom burden will be measured with the IGSQ-13 questionnaire. The IGSQ-13 is an interviewer-administered questionnaire which measures how well the infant tolerates his/her feedings from the parent's/caregiver's perspective. The questionnaire is composed of 13 questions, categorized into 5 symptom domains of stooling, vomiting/spitting-up, crying, fuzziness, and flatulence and summed to calculate an index score.
Changes in Weight from baseline to 57 days | Study Day 57, corresponding to infant age of 78-85 days
  weight (kg)
Changes in Length from baseline to 57 days | Study Day 57, corresponding to infant age of 78-85 days
  length (cm)
Changes in Head Circumference from baseline to 57 days | Study Day 57, corresponding to infant age of 78-85 days
  head circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira M Estorninos, Principal Investigator — University of Alberta
Locations (1):
- Asian Hospital and Medical Center, City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Undecided